CLINICAL TRIAL: NCT00394511
Title: Phase III Randomized Evaluation of Adjuvant Radiotherapy vs No Adjuvant Therapy Following Radical Prostatectomy and Pelvic Lymphadenectomy in Surgical Stage C Adenocarcinoma of the Prostate
Brief Title: Radiation Therapy After Prostatectomy in Treating Patients With Stage III Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: SWOG Cancer Research Network (Network); NCIC Clinical Trials Group (Network); Cancer and Leukemia Group B (Network); Eastern Cooperative Oncology Group (Network); North Central Cancer Treatment Group (Network); Radiation Therapy Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02483; SWOG-8794; CAN-NCIC-PR2; CLB-9493; EST-9887; NCCTG-895251; RTOG-9019; INT-0086; CDR0000075112 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2006-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (2):
- Arm I (Experimental): Radiotherapy. Irradiation of the prostatic bed using megavoltage equipment with effective photon energies of greater than 4 MV.
  Interventions: Procedure: low-LET photon therapy
- Arm II (No Intervention): No further treatment.

INTERVENTIONS:
Procedure: low-LET photon therapy
  Arms: Arm I

SUMMARY:
Randomized phase III trial to compare treatment with or without adjuvant radiation therapy in men with stage III prostate cancer who have had radical prostatectomy and lymphadenectomy recently. Radiation therapy uses high-energy x-rays to damage tumor cells and may be an effective treatment for prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Compare disease-free survival rates of patients randomly assigned to adjuvant external-beam radiotherapy vs. no adjuvant therapy following radical prostatectomy and pelvic lymphadenectomy for surgical Stage C (T3 N0 M0) adenocarcinoma of the prostate.

II. Determine the qualitative and quantitative toxicities associated with this adjuvant therapy.

OUTLINE: Randomized study. Randomization takes place when the patient is physically able to begin treatment, any time within 16 weeks after surgery.

Arm I: Radiotherapy. Irradiation of the prostatic bed using megavoltage equipment with effective photon energies of greater than 4 MV.

Arm II: No further treatment.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Pathologically documented Stage C (T3 N0 M0) adenocarcinoma of the prostate following radical prostatectomy and pelvic lymphadenectomy for clinical Stage A/B disease
* Ineligible for SWOG protocols of higher priority
* At least 1 of the following on pathologic examination:

  * Presence of cancer in the seminal vesicles
  * Evidence of cancer at the inked surgical margin of the prostate
  * Extension of tumor beyond the prostatic capsule
* Negative preoperative metastatic survey within 6 months prior to registration, including the following:

  * Normal bone scan
  * No palpable evidence of extraprostatic tumor extension
* Bilateral lymph node dissection histologically negative for cancer
* Nodal sampling not required with the following stage/biopsy specimen Gleason score/preoperative PSA:

  * Stage T1a/2-6/<10 ng/ml
  * Stage T1b-c/2-5/<10 ng/ml
  * Stage T2a/2-6/<10 ng/ml
  * Stage T2b/2-6/<6 ng/ml
  * Stage T2c/2-6/<4 ng/ml
* Free from the following postoperative complications:

  * Total urinary incontinence
  * Intraoperative rectal injury
  * persistent urinary extravasation
  * Pelvic infection
* Concurrent registration on protocol SWOG-9205 (serum repository protocol) optional
* Concurrent registration on protocol SWOG-8994 (quality-of-life study) required of English-speaking and Spanish-speaking patients enrolled by SWOG

--Patient Characteristics--

* Age: Any age
* Performance status: SWOG 0-2
* Life expectancy: At least 2 years
* Hematopoietic:

  * WBC at least institutional LLN
  * Platelets at least institutional LLN
* Hepatic: SGOT no more than 2 x ULN
* Other: No second malignancy within 5 years except adequately treated nonmelanomatous skin cancer

--Prior Concurrent Therapy--

* Chemotherapy: No prior chemotherapy for prostate cancer
* Endocrine therapy: No more than 3 months of hormonal therapy prior to prostatectomy allowed
* Radiotherapy: No prior radiotherapy for prostate cancer
* Surgery: Radical prostatectomy and pelvic lymphadenectomy within 16 weeks prior to registration required

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 1988-08; Primary Completion 2006-12 (Actual)

REFERENCES:
- [Background] Thompson IM, Paradelo JC, Crawford ED, Coltman CA, Blumenstein B. An opportunity to determine optimal treatment of pT3 prostate cancer: the window may be closing. Urology. 1994 Dec;44(6):804-11. doi: 10.1016/s0090-4295(94)80161-4. No abstract available. PMID 7985307
- [Result] Swanson GP, Thompson IM, Tangem C, et al.: Phase III randomized study of adjuvant radiation therapy versus observation in patients with pathologic T3 prostate cancer (SWOG 8794). [Abstract] Int J Radiat Oncol Biol Phys 63 (Suppl 1): A-1, S1, 2005.
- [Derived] Thompson IM Jr, Tangen CM, Paradelo J, Lucia MS, Miller G, Troyer D, Messing E, Forman J, Chin J, Swanson G, Canby-Hagino E, Crawford ED. Adjuvant radiotherapy for pathologically advanced prostate cancer: a randomized clinical trial. JAMA. 2006 Nov 15;296(19):2329-35. doi: 10.1001/jama.296.19.2329. PMID 17105795